CLINICAL TRIAL: NCT02439554
Title: Risk Factors for Medium-term Adverse Outcomes and Predictive Modeling for Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, Susana García Gutiérrez, PhD, Md, Hospital Galdakao-Usansolo
Other Study IDs: PI12/01842
Record Dates: First submitted 2015-05-04; First posted 2015-05-08 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This subproject is included in a project coordinated between program groups Evaluation of Health Services of Epidemiology and Public Health (Project CAMISS). The overall objective is to evaluate different aspects of health care received by patients with breast cancer from the diagnostic process, treatment, complications, survival and quality of life, to provide information to improve the effectiveness of interventions, reduce variability, have best predictive rules and increase the quality of life. The main objective of the subproject is to create and validate prospectively predictive rules of recurrence, complications, mortality, changes in quality of life in these patients at admission and one/two years of treatment and to evaluate the external validity of our rules to predict relapses, complications and mortality in the retrospective sample of patients participating in screening programs. Observational methodology with information available from a retrospective cohort of women diagnosed between 2000 and 2009 and another 2-year prospective follow-up included 2040 incident cases of breast cancer in 18 hospitals of 5 regions. Cohorts will learn clinical and health care diagnosis, tumor, treatment, hospital, follow-up (complications, relapse, and vital status) cost and quality of life. Prediction rules are created by means of regression/Cox models at the prospective sample and also investigators will assess the external validity in the retrospective cohort in the case of recurrence, complications and mortality. Expected results: There are currently no results of cohort analysis of the diagnostic process of care that integrates different aspects. The study will create tools to assist prognostic and therapeutic decision making process in these patients

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 with both incidental in situ and infiltrating breast cancer.

Exclusion Criteria:

* Lymphoma, sarcoma, lobular carcinoma in situ and inflammatory carcinoma of the breast are excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with both in situ and infiltrating breast cancer
Sampling Method: Probability Sample
Enrollment: 1463 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in quality of life questionnaire module for breast cancer patients | Change from baseline in quality of life at 2 years

SECONDARY OUTCOMES:
Mortality data | Mortality at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susana GArcía, PhD, MD, Principal Investigator — Hospital Galdakao-Usansolo
Locations (1):
- Hospital Galdakao-Usansolo, Galdakao, Bizkaia, Spain

REFERENCES:
- [Derived] Garcia-Gutierrez S, Orive M, Sarasqueta C, Legarreta MJ, Gonzalez N, Redondo M, Rivero A, Serrano-Aguilar P, Castells X, Quintana JM, Sala M; REDISSEC-CaMISS group. Health services research in patients with breast cancer (CAMISS-prospective): study protocol for an observational prospective study. BMC Cancer. 2018 Jan 8;18(1):54. doi: 10.1186/s12885-017-3926-9. PMID 29310641